CLINICAL TRIAL: NCT04021615
Title: Comprehensive Rehabilitation Program Versus Traditional Chest Physiotherapy for Weaning From Mechanical Ventilator
Brief Title: Rehabilitation Program for Weaning From Mechanical Ventilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherin Hassan Mohammed Mehani (Other)
Responsible Party: Sponsor-Investigator, Sherin Hassan Mohammed Mehani, Chairman of Physical Therapy Department of Internal Medicine and Vic Dean for Education and Student Affairs , Faculty of Physical Therapy , Beni- Suef University, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/05032019/ELMoutaz
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-07

CONDITIONS: Mechanical Ventilation Complication
Keywords: rehabilitation; general surgery; difficult weaning

STUDY DESIGN:
Intervention Model Description: Fifty general surgery patients who are difficult and prolonged weaning patients from both sexes (men & women) with age ranged from 40 to 50 years old in surgical intensive care unit, Kasr Al Ainy Teaching Hospital, Cairo University and Beni- Suef Teaching Hospital , Beni -Suef University.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (study group) (Experimental): Twenty five patients will receive comprehensive rehabilitation program combined with inspiratory muscle training.
  Interventions: Other: Comprehensive physical therapy rehabilitation program combined with inspiratory muscle training
- Group B (Control group) (Active Comparator): Twenty five patients will receive traditional chest physical therapy combined with inspiratory muscle training.
  Interventions: Other: Traditional chest physical therapy rehabilitation program combined with inspiratory muscle training

INTERVENTIONS:
Other: Comprehensive physical therapy rehabilitation program combined with inspiratory muscle training — A threshold inspiratory muscle trainer will be connected to the artificial airway with 15 mm and 22 mm adaptors. Training bouts consist of three to five sets of six repetitions breathing through the trainer. Training will be conducted with the patient in bed with an approximately 30° head-up tilt and with intensity about 40 %- 50 % of maximal inspiratory pressure. Patients will be returned to mechanical ventilation for rest between training sets as needed. Three to five sets of six training breaths will be completed for a total of 18 to 30 training breaths per session. Following each training set, the patient indicated a rating of perceived inspiratory exertion on modified Borg scale . The study group will also receive comprehensive rehabilitation program consist of upper-extremity exercises, lower extremity exercises, pedaling exercises, trunk control exercises and bedside functional training
  Other Names: Comprehensive physical therapy rehabilitation program
  Arms: Group A (study group)
Other: Traditional chest physical therapy rehabilitation program combined with inspiratory muscle training — The same inspiratory muscle training for the study group combined with the traditional physical therapy program consist of positioning , modified postural drainage , percussion , vibration.
  Other Names: Traditional physical therapy rehabilitation program
  Arms: Group B (Control group)

SUMMARY:
Statement of the problem:

Are there any differences between comprehensive rehabilitation program consisted of (peripheral muscle training and functional training) combined with inspiratory muscle training and traditional chest physical therapy consisted of (percussion, mechanical vibration, positioning and modified postural drainage) combined with inspiratory muscle training on weaning from mechanical ventilation as a primary outcome, respiratory muscle strength, peripheral muscle strength and functional status in difficult and prolonged weaning from mechanical ventilation as secondary outcomes?

Purpose of the study:

The aim of the present study will be to compare between the effect of comprehensive rehabilitation program combined with inspiratory muscle training and traditional chest physical therapy combined with inspiratory muscle training on weaning from mechanical ventilation as a primary outcome, inspiratory muscle strength, peripheral muscle strength, functional status as secondary outcomes.

DETAILED DESCRIPTION:
Significance of the study Survival of critically ill patients has increased as a result of medical technology and interdisciplinary team cooperation.

Functional losses , reduced quality of life and survival , and increased healthcare costs are consequences of prolonged immobility in ICU.

The European Respiratory Society and European Society of Intensive Care Medicine task force has recommended a hierarchy of ICU mobilization based on progressively increasing exercise intensity; decubitus change and functional positioning , passive mobilization , active- assisted and active exertion , cycloegonometry in bed , sitting in bed orthostatism , static walking , transferring from bed to chair, chair exertion and walking.

Failure to wean may have different etiologies such as underlying severe respiratory disease, respiratory muscle dysfunction , metabolic and endocrine disorders and cognitive dysfunction. Peripheral and respiratory muscles dysfunction is a consequence of prolonged mechanical ventilation and ICU- acquired weakness. Weaning from mechanical ventilator should be considered to be as early as possible to avoid complications caused by absence of spontaneous breathing and further muscles atrophy.

Targeted mobility therapy (TMT) , simulating comprehensive rehabilitation program that will be used in the present study, is a novel strategy for managing critically ill patients . This concept will work as a scientifically- driven, dynamic bundle of rehabilitation intervention that include inspiratory muscle strength training , bronchial hygiene , and active mobilization . This concept will guarantee the bet outcomes for critically ill patients with difficult and prolonged weaning as regards weaning success , days on mechanical ventilator , length of hospital stay and functional mobility.

ELIGIBILITY:
Inclusion Criteria:

* The general surgery patients who fail one weaning attempt of spontaneous breathing trial
* Conscious patients
* Hemodynamically stable patients (lack of hypotension or a need for only low-dose pressors)
* The patients with Acute Physiology and Chronic Health Evaluation II (APACHE II) scale 20 or less

Exclusion Criteria:

* patients with persistent altered sensorium
* patients with major cardiac arrhythmia
* patients with comorbid medical conditions (e.g., neurological diseases) or who are under any sedative or paralytic agents that would interfere with strength measurements and limb exercises
* patients with history of underlying neuromuscular disease or acquired polyneuromyopathies
* patients who are unable to perform physical training due to preexisting joint dysfunction
* obese patients

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-21 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
percentage of successful weaning in both groups | 30 days maximum or until extubation
  Spontaneous breathing trials will be used when underlying cause of acute respiratory failure stabilizes or significantly improves and daily assessment of the patient's readiness for ventilator discontinuation is considered. The spontaneous breathing trial will last from 30 minutes to 120 minutes combined with CPAP and if the trial had failed, the patient will be returned back to full ventilatory support for at least 24 hours before performing a new trial Weaning success is defined as extubation and the absence of ventilatory support 48 hous following extubation
inspiratory muscle strength (MIP) | 30 days maximum or until extubation
  The mechanical ventilator will be used to measure the plateau pressure (maximal inspiratory pressure). Plateau pressure was measured using the inspiratory hold function on the venilator while the patient will be sedated and on volume control mode (Sidebotham et al., 2007) The plateau pressure will be measured by ventilator in millibar then it converted to cm o by multiplying it by 1.01971621298 (1millibar equals 1.01971621298 cm 0) and near the figure to the nearest two decimal places

SECONDARY OUTCOMES:
Upper and lower extremity muscle strength | 30 days maximum or until extubation from mechanical ventilator successfully
  Upper and lower extremity muscle strength will be assessed using a handheld dynamometer. The shoulder flexor, elbow flexor, and knee extensor muscle groups w ill be included in the measurements. Standard test positions will be modified because all patients in this study are using mechanical ventilator and unable to sit up at initial examination. The shoulder and elbow flexors will be tested in the semi-Fowler position. The isometric force of the shoulder flexors will be tested with the shoulder flexed 90 degrees and the elbow in extended position. The dynamometer will be placed just proximal to the epicondyles of the humerus, and the patients will be stabilized at the axillary region. The isometric force of the elbow flexors will be tested with the elbow flexed 90 degrees, the forearm supinated, and the shoulder in neutral position; the dynamometer will be placed just proximal to styloid processes of ulna and radius, and the patients will be stabilized at the superior aspect of
The Functional Independence Measure (FIM) | 30 days maximum or until extubation
  5 activities with The Functional Independence Measure (FIM) were measured, which are bathing, dressing, moving from bed to chair, bowel management, and bladder management.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem ELMoutaz, Professor, Study Director — Faculty of Medicine , Beni -Suef University
Locations (1):
- surgical intensive care unit, Kasr Al Ainy Teaching Hospital, Cairo University and Beni- Suef Teaching Hospital , Beni -Suef University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Description for inclusion and exclusion criteria , procedure for evaluating outcomes and intervention in details
Supporting Information: Study Protocol
Time Frame: 2 months
Access Criteria: I am willing to share data through my E- mail

REFERENCES:
- [Background] Nava S, Fasano L. Inspiratory muscle training in difficult to wean patients: work it harder, make it better, do it faster, makes us stronger. Crit Care. 2011;15(2):153. doi: 10.1186/cc10125. Epub 2011 Apr 18. PMID 21542873